CLINICAL TRIAL: NCT06186024
Title: A PROSPECTIVE, MULTICENTER, SINGLE-ARM TRIAL FOR THE NEW SIZES OF BRIDGE STENTS FOR VERTEBRAL ARTERY STENOSIS: Bridge-MAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bridge-2023-01-1A
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Brain Diseases; Vertebral Artery Thrombosis; Vertebral Artery Stenosis
MeSH Terms: conditions — Brain Diseases; Vertebrobasilar Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Bridge
  Interventions: Device: Bridge

INTERVENTIONS:
Device: Bridge — Stent implantation

SUMMARY:
Aprospective, multicentre, single-arm clinical trial in which approximately 36 subjects would be enrolled using the Bridge 4.5 mm and 5.0 mm stent in accordance with the inclusion and exclusion criteria in this protocol. The success rate of immediate post-procedure stent target lesion treatment was recorded for all subjects, and the incidence of in-stent restenosis (≥50% stenosis) was assessed by DSA imaging follow-up at 6 months (±30 days) post-procedure. The subjects were also followed up at 30 days (±7 days), 6 months (±30 days), and 12 months (±60 days) after stent implantation to assess safety events during the follow-up period. .

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above (including 18 years old), 80 years old below (including 80 years old), male or women with pregnancy test (-); 2. Symptomatic vertebral artery stenosis patients who have failed in medical treatment (defined as patients who have suffered from stroke or TIA within 90 days, and are taking at least one antithrombotic drugs as well as interventions in other vascular risks, such as hypertension and hyperlipidemia decompression or lipid reducing); 3. DSA angiography showed target lesion stenosis degree ≥70% (Stenosis degrees are determined according to WASID method); 4. Diameter of normal blood vessels distal to the target lesion ≥3.5mm and the length of target lesion ≤23mm; 5. Modified Rankin score <3; 6. Patients who are suitable for implantation of rapamycin target eluting vertebral artery stent and are voluntary to

Exclusion Criteria:

* Presence of tandem stenotic lesions (≥50% tandem stenosis) in the target lesion area; (2) TIA or non-disabling stroke due to factors other than vertebral artery stenosis (e.g. atrial fibrillation, etc.); (3) Previous surgical treatment or endovascular intervention in the target lesion area; (4) Comorbid severe systemic systemic diseases or other diseases with a potential risk of sudden death, or subjects with a life expectancy of <1 year; (5) Subjects with contraindications to heparin, aspirin, clopidogrel, or other antiplatelet drugs and who cannot tolerate anticoagulant and antiplatelet drug therapy; (6) Previous cerebral infarction with residual responsible vascular-related severe neurological deficits (mRS ≥3 points); (7) Previous severe myocardial infarction within 2 weeks; (8) Accompanied by other intracranial lesions such as intracranial haemorrhage, aneurysm, arteriovenous malformation, intracranial tumour, etc (9) Non-atherosclerotic stenosis such as arterial entrapment, smoker's disease, active arteritis, and unknown causes; (10) Severe tortuosity or calcification of the target vessel that precludes implantation of a stent or lesion that cannot be dilated; (11) Severe renal impairment, or those who are allergic or resistant to contrast agents, rapamycin (Rapamycin) and its derivatives, cobalt-based alloys, PDLLA; (12) Pregnant or lactating women; (13) Patients participating in other drug or device studies that have not met endpoints

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of in-stent restenosis at 6 months postoperatively | 180±30 days

SECONDARY OUTCOMES:
Technical Success | post-implantation immediately
  DSA suggesting residual stenosis ≤20% after implantation
Any death or stroke during the follow-up associated with treatment in the target vessel supply region | 1 year after stent implantation
  Number of participants with death or stroke related to treatments for target vessel blood supply area
Any death or stroke | 1 year after stent implantation
  Number of participants with death or stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Affilicated to Captical Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided